CLINICAL TRIAL: NCT06119646
Title: The Effect of Warm Pads Applied to the Breast During Episiotomy Repair on the Amount of Milk, Breastfeeding Motivation and the Perception of Insufficient Milk
Brief Title: Warm Pads Applied to the Breast During Episiotomy Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: Lansinoh Laboratories (Industry)
Responsible Party: Principal Investigator, Asiye Tutca, Midwifery, Student of Master, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 223278001012
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Breastfeeding
Keywords: warm pads; perception of insufficient milk
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm Pads Applied to the Breast (Experimental): When repairing the episiotomy of a pregnant woman who has given birth, a pad heated in a microwave oven at 180 W for 1 minute is applied to each breast for 20 minutes. The application is made when the temperature of the pad, measured with a thermometer, reaches a maximum of 40.5 C.
  Interventions: Other: Warm Pads Applied to the Breast
- Control (No Intervention): A routine care was performed.

INTERVENTIONS:
Other: Warm Pads Applied to the Breast — Applying a warm pad to a breast during episiotomy repair
  Arms: Warm Pads Applied to the Breast

SUMMARY:
H1-1 Hypothesis: Warm pads applied to the breast during episiotomy repair in the intervention group will have an effect on increasing milk production compared with the control group.

H1-2 Hypothesis: Warm pads applied to the breast of the intervention group during episiotomy repair will have an effect on increasing breastfeeding motivation compared to the control group.

H1-3 Hypothesis: Warm pads applied to the breast of the intervention group during episiotomy repair will have an effect on reducing the mother's perception of insufficient milk compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* First pregnancy,
* Those who are 18 years or older,
* Can speak Turkish and express themselves in Turkish,
* Do not have any disability (such as sight, hearing),
* Gave birth after >37 weeks of pregnancy,
* Who have had a normal birth and have had an episiotomy,
* There is no open wound on the breast,
* A singleton pregnancy,
* Women who are open to communication and mentally and emotionally healthy.

Exclusion Criteria:

* Those who do not agree to work
* Those who want to leave for any reason during the application process
* Having postpartum haemorrhage,
* Women who develop any postpartum complications,
* Women whose babies are admitted to the neonatal intensive care unit.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | pre-intervention
  The Introductory Information Form is a 15-item survey form prepared by researchers based on the literature. The Introductory Information Form includes 10 questions on socio-demographic characteristics of pregnant women and their partners and 5 questions on obstetric characteristics of pregnant women.
Postpartum Milk Expression and Amount Information Form | in the first hour in postpartum period
  Postpartum Milk Expression and Amount Information Form aims to be evaluated by researchers by asking 8 questions to the intervention group and 6 questions to the control group. The questions were prepared by the researcher. There are statements that need to be measured quantitatively and recorded by the researcher.

SECONDARY OUTCOMES:
Primiparous Breastfeeding Motivation Scale (PBMS) | in the second hour in postpartum period
  The scale, whose Turkish validity and reliability was confirmed by Akçay and Demirgöz Bal in 2019, was published by Stockdale et al. in 2013. PBMS is a 37-item scale developed to evaluate the postnatal breastfeeding motivation in primipara. The scale has four sub-dimensions of "The value placed on breastfeeding", "Self-efficacy", "Perceived support from the midwife" and "Expectation of success". High scores from the scale indicate high breastfeeding motivation, low scores indicate low breastfeeding motivation.
Perception of Insufficient Milk Supply Questionaire | in the second hour in postpartum period
  The scale, developed by McCarter-Spaulding and Kearney in 2001, consists of 6 questions to determine the perception of insufficient breast milk. The Turkish validity and reliability of the scale was conducted by Gökçeoğlu and Küçükoğlu in 2014. The first question of the scale asks whether the mother feels that her milk is sufficient, and is answered with 'yes' or 'no'. Other questions on the scale aim to measure the perception of milk inadequacy. These questions are scored on a scale from 0 to 10 ('0' means the milk is perceived as completely inadequate, '10' means the milk is perceived as completely sufficient). The scale can produce scores from 0 to 50, and a higher total score indicates an increasing perception of milk adequacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Faculty of Medicine Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting in June 2024
Access Criteria: IPD data will be shared with the principal investigator.

REFERENCES:
- [Result] An official position statement of the Association of Women's Health, Obstetric and Neonatal Nurses. Breastfeeding and the Use of Human Milk. Nurs Womens Health. 2021 Oct;25(5):e4-e8. doi: 10.1016/j.nwh.2021.06.005. Epub 2021 Jul 22. No abstract available. PMID 34305016
- [Result] Gökçeoğlu, E. ve Küçükoğlu, S. (2018). Validity and Reliability Study of Perception of Insufficient Milk Supply Questionnaire for Turkish Society. International Journal of Innovative Research and Reviews, 2(2), 15-20.
- [Result] Lin, L. ve Zhang, T. (2011). Playing exergames in the classroom: Pre-service teachers' motivation, passion, effort, and perspectives. JTATE, 19(3), 243-260.
- [Result] McCarter-Spaulding DE, Kearney MH. Parenting self-efficacy and perception of insufficient breast milk. J Obstet Gynecol Neonatal Nurs. 2001 Sep-Oct;30(5):515-22. doi: 10.1111/j.1552-6909.2001.tb01571.x. PMID 11572532
- [Result] Ryan RM, Deci EL. Intrinsic and Extrinsic Motivations: Classic Definitions and New Directions. Contemp Educ Psychol. 2000 Jan;25(1):54-67. doi: 10.1006/ceps.1999.1020. PMID 10620381
- [Result] Saus-Ortega C. Promoting correct positioning and attachment in breastfeeding infants born by section cesarean in the La Fe Hospital in Spain: a best-practice implementation project. JBI Evid Implement. 2020 Sep;18(3):297-307. doi: 10.1097/XEB.0000000000000230. PMID 32516210
- [Result] Stockdale J, Sinclair M, Kernohan G, McCrum-Gardner E, Keller J. Sensitivity of the breastfeeding motivational measurement scale: a known group analysis of first time mothers. PLoS One. 2013 Dec 31;8(12):e82976. doi: 10.1371/journal.pone.0082976. eCollection 2013. PMID 24391731